CLINICAL TRIAL: NCT03552263
Title: A Double-blind, Randomized and Placebo-controlled Phase 2 Study to Evaluate the Safety and Efficacy of T89 in Prevention and Treatment of Acute Mountain Sickness (AMS) During Rapid Ascent
Brief Title: Safety and Efficacy of T89 in Prevention and Treatment of Adults With Acute Mountain Sickness (AMS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tasly Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T89-30-AMS; NCT03621410 (obsolete NCT alias)
Record Dates: First submitted 2018-05-25; First posted 2018-06-11 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Acute Mountain Sickness (AMS)
Keywords: Acute mountain sickness
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Intervention Model Description: This study is a prospective, double-blind, randomized, placebo-controlled phase 2 clinical trial having three arms including T89 low-dose, T89 high-dose and a placebo controlled group. People will be screened against the inclusion/exclusion criteria after informed consent. Eligible subjects will be randomly assigned into one of three arms and instructed to use T89 orally twice daily for 14 days (Days 1-14) before ascending, and 5 days after ascending during the observation period (Days 15-19). Specifically, for subjects in the T89 high-dose group, they will take placebo instead of T89 from Day 1 to Day 12, and take T89 on Days 13-14. The primary efficacy parameter is Lake Louise Scoring System (LLSS) which will be evaluated by subject-self and principal investigator in clinic. Other efficacy parameters include Visual Analog Scales (VAS), exercise tolerance, blood lactate, and blood oxygen saturation that will be performed at altitude.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- T89 low-dose group (Experimental): T89 capsule is a botanical drug containing 75mg active substance which is the water extract of Danshen and Sanqi. Placebo capsule does not contain any amount of active substance.
  Subjects in this group will use three T89 capsules and one Placebo capsule each time by oral administration twice daily for 19 days.
  Interventions: Drug: T89 capsule; Drug: Placebo capsule
- T89 high-dose group (Experimental): T89 capsule is a botanical drug containing 75mg active substance which is the water extract of Danshen and Sanqi. Placebo capsule does not contain any amount of active substance.
  Subjects in this group will use four Placebo capsules each time by oral administration twice daily for 12 days followed by using four T89 capsules each time by oral administration twice daily for 7 days
  Interventions: Drug: T89 capsule; Drug: Placebo capsule
- Placebo group (Placebo Comparator): Placebo capsule does not contain any amount of active substance. Subjects in this group will use four Placebo capsules each time by oral administration twice daily for 19 days.
  Interventions: Drug: Placebo capsule

INTERVENTIONS:
Drug: T89 capsule — T89 capsules (75mg), orally, twice daily.
  Arms: T89 high-dose group; T89 low-dose group
Drug: Placebo capsule — Placebo capsules (0mg), orally, twice daily.

SUMMARY:
Acute mountain sickness (AMS) is one of three syndromes of altitude illness. It is very common when people venture over 2500 meters altitude. This illness is mainly induced by acute exposure to low partial pressure of oxygen at high altitude that will cause a pathological effect on humans. T89 capsule is a modernized industrialized traditional Chinese herbal medicine. It is a botanical drug for oral use. In recent years, several literatures and clinical studies have showed that oral administration of T89 may provide substantial benefits in the prevention or alleviation of symptoms associated with acute mountain sickness (AMS), including nausea, vomiting, headache, dizziness, fatigue, and sleep disturbance. Such effect was also observed in a pilot clinical study recently conducted in Tibet in China.

This study is a prospective, double-blind, randomized, placebo-controlled phase 2 clinical trial having three arms including T89 low-dose, T89 high-dose and a placebo controlled group. People will be screened against the inclusion/exclusion criteria after informed consent signed. Eligible subjects will be randomly assigned into one of three arms and instructed to use T89 orally twice daily for 14 days (Days 1-14) before ascending, and 5 days after ascending during the observation period (Days 15-19). The primary efficacy parameter is Lake Louise Scoring System (LLSS) which will be evaluated by subject-self and principal investigator in clinic.

DETAILED DESCRIPTION:
Acute mountain sickness (AMS) is one of three syndromes of altitude illness. It is very common when people venture over 2500 meters altitude. This illness is mainly induced by acute exposure to low partial pressure of oxygen at high altitude that will cause a pathological effect on humans. It presents a syndrome characterized by a collection of nonspecific symptoms, including headache and one of the following: gastrointestinal symptoms, fatigue and/or weakness, dizziness/light headedness or difficulty sleeping. Severity and incidence of these symptoms depend on the speed of ascent, altitude, duration of altitude exposure, physical exertion, and inherent genetic susceptibility.

T89 capsule is a modernized industrialized traditional Chinese herbal medicine. It is a botanical drug for oral use. The active substance is the water extract of Danshen (Radix Salivae Miltiorrhizae, RSM) and Sanqi (Radix Notoginseng, RN). T89 capsule also contains Bingpian (Borneol) which may promote absorption of the active substance. In recent years, several literatures and clinical studies have showed that oral administration of T89 may provide substantial benefits in the prevention or alleviation of symptoms associated with acute mountain sickness (AMS), including nausea, vomiting, headache, dizziness, fatigue, and sleep disturbance. Such effect was also observed in a pilot clinical study recently conducted in Tibet in China.

This study is a prospective, double-blind, randomized, placebo-controlled phase 2 clinical trial having three arms including T89 low-dose, T89 high-dose and a placebo controlled group. People will be screened against the inclusion/exclusion criteria after informed consent signed. Eligible subjects will be randomly assigned into one of three arms and instructed to use T89 orally twice daily for 14 days (Days 1-14) before ascending, and 5 days after ascending during the observation period (Days 15-19). Specifically, for subjects in the T89 high-dose group, they will take placebo instead of T89 from Day 1 to Day 12, and take T89 on Days 13-14. The primary efficacy parameter is Lake Louise Scoring System (LLSS) which will be evaluated by subject-self and principal investigator in clinic. Other efficacy parameters include Visual Analog Scales (VAS), exercise tolerance, blood lactate, and blood oxygen saturation that will be performed at altitude. The primary efficacy endpoint is the difference in LLSS total scores on Day 16 morning (12 hours after arrival at high altitude) compared between T89 and Placebo group. A total of 120 subjects will be enrolled with approximately 40 subjects in each arm, and a minimum of 100 subjects are expected to complete the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers: ages 18 - 55 years old;
2. Primary residence elevation of 1,000 ft or lower;
3. Not ascending to altitude >10,000 ft within 4 months prior to screening;
4. Females of childbearing potential must have a negative pregnancy test, not be breast feeding and established on a method of contraception that in the investigator's opinion is acceptable. Females must agree to remain on their established method of contraception from the time of the screening visit and throughout the study period.
5. Willing to participate voluntarily and to sign a written informed consent.

Exclusion Criteria:

1. Subjects with medical history of cardiovascular, cerebrovascular diseases or asthma;
2. Subjects with clinically significant respiratory system disease, digestive disease, mental disease, metabolic disease, acute infection or anemia;
3. Total LLSS self-assessment score and clinical assessment score is greater than 1 before ascending (Screening visit and Visit 1);
4. Blood oxygen saturation (SpO2) <95% at sea level;
5. Subjects with abnormal renal or liver function with clinical significance (alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2×upper limits of normal(ULN), Creatinine> ULN);
6. Subjects with C reactive protein (CRP) > ULN;
7. Subjects with primary headache;
8. Surgery or blood donation within 3 months prior to screening;
9. On treatment of any medications (including any dietary supplements)except for birth control within 14 days prior to screening and throughout the study period;
10. Contradictive to treatment of Danshen (Radix Salivae Miltiorrhizae, RSM) products;
11. Women in pregnancy or lactation period;
12. Substance abuse. Subjects with a recent history (within the last 2 years) of alcoholism or known drug dependence;
13. Participation in any other clinical trial or on an investigational drug within 30 days prior to screening;
14. A family member or relative of the study site staff;
15. Any other condition that, in the opinion of the investigator, is likely to prevent compliance with the study protocol, interfere with the assessment, or pose a safety concern if the subject participates in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2019-10-20 (Actual); Study Completion 2019-11-10 (Actual)

PRIMARY OUTCOMES:
The LLSS self- and clinical assessments score on Day 16 morning(next morning of arrival at high altitude) between T89 and Placebo groups. | Day 16 morning (next morning of arrival at high altitude)
  Lake Louise Scoring System (LLSS) self-assessment score [0-15]. Lake Louise Scoring System (LLSS) clinical assessment score [0-10]. Lake Louise Scoring System (LLSS) self-and clinical assessment score [0-25].The higher LLSS score, the worse symptoms of AMS. The Lake Louise Scoring System (LLSS) will be assessed by subject-self and clinic staff (principal investigator or sub- investigator) twice daily from Day 15 to Day 19. And the difference in LLSS total scores on Day 16 morning (next morning of arrival at high altitude) is pre-specified as primary efficacy endpoint compared between T89 and Placebo groups.

SECONDARY OUTCOMES:
The area under the curve (AUC) of LLSS self- and clinical assessments score in the mean LLSS score-time profile during rapid ascent (Days 15-19) between T89 and Placebo groups. | Day 15 to Day 19 after initiation of treatment
  LLSS assessments will be conducted twice per day: before breakfast and before sleep. The area under the curve (AUC) of LLSS total scores in the mean LLSS score-time profile during rapid ascent (Days 15-19) will be compared between T89 and Placebo groups.
The total incidence of AMS evaluated by LLSS between T89 and Placebo groups. | Day 15 to Day 19 after initiation of treatment
  The difference in total incidence of AMS (using LLSS to evaluate) will be compared between T89 and Placebo groups. AMS is defined as: (a) symptom of headache and LLSS self-assessment score ≥2, or (b) symptom of headache and any LLSS score ≥3.
The mean total Visual Analog Scales (VAS) scores of headache during rapid ascent (Days 15-19) between T89 and Placebo groups. | Day 15 to Day 19 after initiation of treatment
  Visual Analog Scales (VAS) scores [0-10]. VAS score of zero (0) represents no pain and VAS score of ten (10) represents the most severe pain (headache) ever.The higher VAS score, the worse pain. VAS scores assessments will be conducted twice per day: before breakfast and before sleep. The difference will be compared in the mean total VAS headache scores during and after rapid ascent from Day15 to Day19 between T89 and Placebo groups.
The exercise tolerance (maximum wattage achieved or watts/kg and difference in watts from sea level to altitude) during rapid ascent (Days 15-19) between T89 and Placebo groups. | Day 15 to Day 19 after initiation of treatment
  The exercise tolerance test will be performed on a computer controlled bicycle ergometer that increases the resistance in steps until the subject is exhausted and stops pedalling. The maximum wattage achieved or watts/kg and difference in watts from sea level to altitude will be compared over Day 15 to Day 19 after rapid ascent between T89 and Placebo groups.
The time from the foot of the mountain to onset of AMS between T89 and Placebo groups. | Day 15 to Day 19 after initiation of treatment
  Subjects will be recorded the time of the first onset of AMS during and after rapid ascent from Day 15 to Day 19. The difference will be compared in time to onset of AMS.
The symptom-related drop-out rate between T89 and Placebo groups. | Day 15 to Day 19 after initiation of treatment
  All dropped-out subjects will be recorded in terms of time of drop-out and reason (s). The "drop-out" over Day 15 to Day 19 as the result of at least one symptom of AMS is pre-defined as symptom-related drop-out, and the difference will be compared in the rate of symptom-related drop-out between T89 and Placebo groups.
The total incidence of progressive diseases (e.g., HAPE, HACE, severe AMS requiring descent or treatment) between T89 and Placebo groups. | Day 15 to Day 19 after initiation of treatment
  All progressive diseases including, but not limited to, high altitude pulmonary adema (HAPE), high altitude cerebral adema (HACE) and severe AMS will be recorded in terms of the start and end time, severity, duration, emergency measurement and outcome over Day 15 to Day 19. The difference will be compared in the total incidence of progressive diseases between T89 and Placebo groups.
The blood oxygen saturation (SpO2) during rapid ascent (Days 15-19) between T89 and Placebo groups. | Day 15 to Day 19 after initiation of treatment
  Blood oxygen saturation (SpO2) will be tested using a pulse oximetry and measured from the left index finger throughout the study. SpO2 will be tested four times daily by site staff before breakfast, before lunch, before dinner, and before sleep from Day 16 to Day 19. But for Day 15, SpO2 will be tested at sea level, arrival at altitude and before sleep. The difference will be compared in SpO2 from sea level to altitude over Day 15 to Day 19 after rapid ascent between T89 and Placebo groups.
The LLSS self- and clinical assessments scores in subjects stratified by pooled median SpO2 value during rapid ascent (Days 15-19) between T89 and Placebo groups. | Day 15 to Day 19 after initiation of treatment
  All subjects will be stratified by comparing individual SpO2 value collected at the corresponding time of LLSS assessment with pooled median SpO2 value. The mean value of LLSS total scores for subjects with value of SpO2 less than pooled median value will be compared between T89 and Placebo groups.
The blood pressure (mmHg) during rapid ascent (Days 15-19) between T89 and Placebo groups. | Day 15 to Day 19 after initiation of treatment
  Unit of blood pressure is mmHg. Both systolic blood pressure (SBP) and diastolic blood pressure (DBP) will be recorded. Blood pressure will be recorded in vital signs from Days 15-19. They will be measured when subject is seated after a 5-min period of inactivity, and the blood pressure is recommended to examine on the same arm throughout the study. The difference will be compared in blood pressure from sea level to altitude over Day 15 to Day 19 after rapid ascent between T89 and Placebo groups.
The heart rate (beats/minute) during rapid ascent (Days 15-19) between T89 and Placebo groups. | Day 15 to Day 19 after initiation of treatment
  Unit of heart rate is beats/minute. Heart rate will be recorded in vital signs from Days 15-19. They will be measured when subject is seated after a 5-min period of inactivity. The difference will be compared in heart rate from sea level to altitude over Day 15 to Day 19 after rapid ascent between T89 and Placebo groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey W Sall, PhD, MD, Principal Investigator — Department of Anesthesia and Perioperative Care, University of California, San Francisco, CA, U.S.
Locations (1):
- Hypoxia Research Lab, UCSF Parnassus Campus, S-256, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No